CLINICAL TRIAL: NCT02639819
Title: A Pilot Study of Ultra-Early Intravenous ɛ-Aminocaproic Acid in Spontanteous Intracerebral Hemorrhage
Brief Title: Management of Intracerebral Hemorrhage With Aminocaproic Acid - Pilot Study
Acronym: MANICHAN-PILOT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn from IRB review on 03/08/16
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160096H
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Stroke; Cerebrovascular
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Aminocaproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Study drug
  Interventions: Drug: ɛ-Aminocaproic Acid

INTERVENTIONS:
Drug: ɛ-Aminocaproic Acid — Intervention: intravenous ε-Aminocaproic Acid within 3 hours of symptom onset
  Other Names: Amicar; Aminocaproic Acid

SUMMARY:
This is single-arm, open-label, safety and feasibility pilot study of ɛ-aminocaproic acid in ICH patients.

Consecutive ICH volume with hematoma volume less than 30 mL by ABC/2 method presenting within 3 hours of symptom onset, meeting all inclusion criteria, and without exclusions will be consented and enrolled. Subjects will receive 5 grams of intravenous ɛ-aminocaproic acid over 1 hour, followed by the same at 1 mg/hour for 23 hours. Comupted tomography (CT) head will be done at 24 hours in order to follow hematoma size. Electrocardiogram, lower extremity venous Doppler and NIHSS will also be done at 24 hours. The patient will be followed in the clinic 30-90 days post discharge for functional status.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Supratentorial ICH ≤ 30 mL in volume and seen on ≥ 2 slices on a 0.5 mm CT head
3. IVH involving < 50% of the ipsilateral lateral ventricle will be allowed
4. Treatment initiated within 1 hour of baseline CT and 3 hours of onset or last known normal

Exclusion Criteria:

1. Baseline mRS ≥ 2
2. Infratentorial hemorrhage (brainstem/cerebellum)
3. Any supratentorial hemorrhage extending to the brainstem
4. ICH > 30 mL
5. Patients who undergo surgical evacuation
6. Presenting outside of the 3 hour window
7. Intraventricular extension > 1/2 of one lateral ventricle
8. Intraventricular extension into the 3rd or 4th ventricle, or the aqueduct or involving >50% of the ipsilateral lateral ventricle
9. ICH due to trauma
10. ICH due to aneurysm of arteriovenous malformation
11. ICH due to underlying neoplasm or infectious mass
12. ICH due to Warfarin or other oral or intravenous anticoagulants
13. International normalization ratio > 1.4
14. Life expectancy < 1 year (prior to ICH onset); due to any cause.
15. History of recent ischemic stroke (within the past 3 months)
16. History of deep vein thrombosis or pulmonary embolism
17. History of recent myocardial infarction (within the past 3 months)
18. Known history of hypercoagulable state
19. History of cancer
20. Glomerular filtration rate < 60 mL/min
21. Received any hemostatic therapy for any indication (last 14 days)
22. Received any investigational therapy in last 90 days
23. "Do Not Resuscitate" order in place or expected, advance directives that could limit aggressive treatment measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hematoma volume | 24 hours
Lower extermity deep vein thrombosis on venous duplex ultrasound | 24-48 hours
Evidence of cardiac ischemia on the electrocardiogram | 24 hours
National Insitutes of Health Stroke Scale score | 24 hours

SECONDARY OUTCOMES:
Modified Rankin Scale score | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Misra, MD, Study Chair — The University of Texas Health Science Center at San Antonio; Jean-Louis Caron, MD, FRCS(C), Study Director — The University of Texas Health Science Center at San Antonio; Reza Behrouz, DO, Principal Investigator — The University of Texas Health Science Center at San Antonio

IPD SHARING:
Plan to Share IPD: No